CLINICAL TRIAL: NCT00546676
Title: A Canadian Multicenter, Prospective, Open Label, Non-Comparative Study of the Effectiveness and Safety of Oral Telithromycin, 800mg Once Daily in the Treatment of Either Community Acquired Pneumonia or Acute Exacerbation of Chronic Bronchitis in Ambulator
Brief Title: Ketek in CAP / AECB in Ambulatory Adult Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMR3647A_4018
Record Dates: First submitted 2007-10-18; First posted 2007-10-19 (Estimated); Last update posted 2007-11-14 (Estimated); Status verified 2007-11

CONDITIONS: Community Acquired Pneumonia (CAP); Acute Exacerbation of Chronic Bronchitis (AECB)
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — telithromycin

INTERVENTIONS:
Drug: Telithromycin

SUMMARY:
To determine the clinical effectiveness of telithromycin in the treatment of either CAP or AECB in a large population of ambulatory adult patients in a community-based setting.

ELIGIBILITY:
Inclusion Criteria:

Male or female subjects greater than or equal to 18 years who fulfill the clinical diagnostic criteria for outpatient treatment of one of the two following community acquired respiratory tract infections (CARTIs):

* CAP: a new pulmonary infiltrate confirmed by chest X-ray and at least 3 of the following signs or symptoms of infection: fever greater than or equal to 38C, cough, chest pain, sputum production, rales, dyspnea, malaise and/or headache; OR
* ECB: documented medical history of chronic bronchitis in subjects over the age of 40 and presenting an FEV1 <80% of the predicted value in the last 36 months and at least 2 of the following clinical symptoms: increased sputum purulence, increased dyspnea and/or increased sputum production.

Exclusion Criteria:

* Subjects with a confirmed cardiogenic syncope, ventricular tachyarrythmia or Torsades de Pointes while taking a medicinal product with QT- prolonging potential, such as a macrolide or quinolone antibiotic, or other non-antibiotic suspected of prolonging the QT interval;
* Pregnancy or lactation;
* Hypersensitivity to macrolides;
* Concomitant treatment with terfenadine, ergot alkaloid derivatives, astemizole or pimozide;
* Myasthenia gravis;
* Antibiotic treatment in the 30 days prior to study entry;
* Treatment with any investigational product in the 30 days prior to study entry and/or a previous participation in this study.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2004-05; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of the clinical effectiveness of telithromycin treatment as determined by the clinical cure rates based on the resolution of infection-related signs and symptoms for CAP and AECB.

SECONDARY OUTCOMES:
Evaluate speed of symptom resolution,define the safety of telithromycin,& assess health economic parameters

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Mississian, Study Director — Sanofi